CLINICAL TRIAL: NCT06574568
Title: A Multicenter, Open-label, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Efficacy of YKST02 in Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of YKST02 in Participants With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Excyte Biopharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YKST02-I-01
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YKST02 (Experimental): Participants will receive different doses of YKST02 in 21-day cycles via intravenous injection.
  Interventions: Drug: YKST02

INTERVENTIONS:
Drug: YKST02 — BCMA-CD3 bispecific antibody
  Other Names: YKST02 for Injection

SUMMARY:
This study aims to provide a basis for further clinical development of YKST02. YKST02 is a study medicine that targets multiple myeloma and activates the human body to fight against this disease.

DETAILED DESCRIPTION:
This study is the first-in-human clinical trial to evaluate the safety, tolerability, pharmacokinetic (PK) profile and preliminary efficacy of YKST02 in patients with relapsed or refractory multiple myeloma (MM). Multiple Myeloma (MM) is a cancer of the blood's plasma cells (blood cell). YKST02 is a bispecific antibody bridging CD3-expressing T cells and BCMA-expressing multiple myeloma cells to induce T cells-mediated cytotoxicity. This study consists of dose escalation phase and dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Participants or their legally acceptable representative must sign an ICF indicating that the participants understand the purpose of, and procedures required for the study and are willing to participate in the study.
2. Diagnosis of multiple myeloma according to the IMWG criteria.
3. Receipt of at least two prior classes of drugs either in separate regimens or as combinations. The three classes are defined as: An immunomodulatory drug, a proteasome inhibitor, and an anti-CD38 drug.
4. Measurable disease at screening, as defined by at least 1 of the following:

   1. Serum M-protein ≥0.5 g/dL;
   2. Urinary M-protein excretion ≥200 mg/24 hours;
   3. Abnormal serum free light chain (FLC) ratio ( <0.26 or >1.65) and serum immunoglobulin FLC≥10 mg/dL.
5. Eastern Cooperative Oncology Group Performance Status (ECOG) of 0-1.
6. An estimated survival time of more than 12 weeks.
7. Recovery to Grade 0-1 (Graded by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0) from adverse events related to prior therapy except alopecia.
8. Adequate hematological and organ function.
9. Female participants of childbearing potential must have a negative serum pregnancy test at screening. Female patients who are sexually active must use highly effective methods of contraception throughout the study and for 3 months following the last dose of study treatment.
10. Male participants must agree to use reliable methods of contraception (barrier methods or sexual abstinence) and avoid sperm donation throughout the study period and until 3 months after the last dose.

Exclusion Criteria:

1. Plasma cell leukemia (>2.0×10^9/L plasma cells by standard differential), Waldenstrom's Macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or primary light-chain amyloidosis.
2. History of antitumor therapy as follows, before the first dose of study drug:

   1. Targeted therapy with small molecule drug within 2 weeks or 5 half-lives, whichever is longer;
   2. Targeted therapy with macromolecular drug or Immunomodulatory agent therapy within 2 weeks;
   3. Chemotherapy within 2 weeks;
   4. Treatment with an investigational drug within 2 weeks or 5 half-lives, whichever is shorter;
   5. Radical/extensive radiotherapy within 4 weeks, or local palliative radiotherapy within 2 weeks, or acute toxicity induced by previous radiotherapy have not recovered to grade ≤1;
   6. Autologous stem cell transplantation within 12 weeks;
   7. History of organ transplant, or allogeneic stem cell transplantation within 6 months;
   8. Prior treatment with any B cell maturation antigen (BCMA) targeted therapy;
   9. Prior treatment with any BCMA targeted chimeric antigen receptor modified [CAR]-T cells therapy.
3. Any active acute graft-versus-host disease (GvHD), grade 2-4 (according to Glucksberg criteria) or active chronic GvHD requiring systemic treatment within 2 weeks.
4. Prior myelodysplastic syndrome or malignancy within 5 years, except for localized malignancies that have been adequately treated or free of the disease for ≥ 5 years, e.g., basal cell carcinoma of the skin, squamous cell carcinoma of the skin, non-muscle invasive bladder cancer, localized prostate cancer, carcinoma in situ of the cervix, carcinoma in situ of the breast.
5. Active central nervous system (CNS) involvement or exhibition of clinical signs of meningeal involvement of multiple myeloma, or other evidence of uncontrolled metastases to the CNS or meninges, judged by the investigator.
6. (a) History of or current relevant CNS pathology as epilepsy, seizure, paresis, aphasia, apoplexia, severe brain injuries, cerebellar disease, organic brain syndrome, psychosis; (b) Evidence for presence of inflammatory lesions and/or vasculitis on cerebral MRI.
7. History or evidence of cardiovascular disease, including:

   1. Acute coronary syndromes (eg, myocardial infarction, unstable angina) within 6 months prior to enrollment;
   2. Coronary angioplasty or stenting within 6 months prior to enrollment;
   3. Clinically significant unstable arrhythmias (eg, atrial fibrillation), however, atrial fibrillation has been controlled for over 30 days prior to the first dose of YKST02 were allowed;
   4. New York Heart Association (NYHA) stage III or higher congestive heart failure within 6 months prior to enrollment; Cardiac valve morphological abnormalities recorded by ECHO (≥ grade 2), note that grade 1 cardiac valve morphological abnormalities (such as mild regurgitation/stenosis) were allowed, but participants with moderate valve thickening were excluded;
   5. Left ventricular ejection fraction (LVEF) below lower limit of the study center, or LVEF<50% if there is no lower limit at the study center;
   6. The Fridericia-corrected QT interval (QTcF) ≥ 470 msec (female) or ≥ 450 msec (male)；
   7. Implantable defibrillator;
   8. Clinically uncontrollable hypertension (i.e., SBP≥160 mm Hg and/or DBP≥100 mm Hg).
8. Known allergy to monoclonal antibody drugs or exogenous immunoglobulin.
9. Any major organ surgery or significant trauma within 4 weeks prior to the first dose of YKST02, or those requiring elective surgeries during the study, and all AEs associated with surgery or significant trauma have not recovered before the first dose of the YKST02.
10. Regular dose of systemic corticosteroids during 4 weeks prior to initiation of study drug, or anticipated need of corticosteroids exceeding prednisone 20 mg/day or equivalent during the trial, or any other systemic immunosuppressive therapy within 4 weeks prior to study entry.
11. Virological tests: Hepatitis B virus surface antigen (HBsAg) positive and/or hepatitis B core antibody (HBcAb) positive, and hepatitis B virus (HBV) deoxyribonucleic acid (DNA) quantitative >ULN of the testing institution; Hepatitis C antibody (HCV-Ab) positive and hepatitis C virus-RNA (HCV-RNA) quantitative > ULN of the testing institution; Anti-human immunodeficiency virus (Anti-HIV) positive. Participants will be excluded from the study if any of the above criteria is met.
12. Uncontrolled active infections requiring oral or intravenous systemic therapy, except for local treatment.
13. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (once a month or more frequently).
14. Pregnant or lactating women.
15. Known mental disorder that may affect study compliance or poor compliance.
16. Receipt of any live attenuated vaccines or live virus vaccine within 4 weeks prior to the first dose of study treatment.
17. Other serious systemic diseases or laboratory abnormalities or other reasons that the investigator believes are not appropriate for participating the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLT) | 21 days after the first dose
  The Dose Limiting Toxicities (DLTs) are based on drug related adverse events and are specifically defined in study protocol.
Incidence of Adverse Events (AEs) | up to 42 weeks
  An AE is defined as any untoward medical event that occurs after a subject receives the investigational drug, which may be manifested as symptoms, signs, diseases, or laboratory abnormalities, but may not necessarily have a causal relationship with the investigational drug.
Incidence of Serious Adverse Events (SAEs) | up to 42 weeks
  A SAE refers to an untoward medical occurrence such as death, life-threatening event, permanent or serious disability or loss of function, need for hospitalization or prolongation of hospitalization after the subject receives the investigational drug, and congenital abnormalities or birth defects.
Overall Response Rate (ORR) | From the date of dosing until the date of first documented progression
  Measured by IMWG criteria, only applicable in dose expansion phase

SECONDARY OUTCOMES:
Area under the Concentration-time Curve (AUC) after Administration | up to 42 weeks
  AUC of YKST02
Maximum Serum Concentration (Cmax) of YKST02 | up to 42 weeks
  Cmax is defined as the maximum observed serum concentration of YKST02
Time to Cmax of YKST02 (Tmax) | up to 42 weeks
  Time to maximum serum concentration (Tmax) of YKST02
Terminal Half-life (T1/2) of YKST02 | up to 42 weeks
  Terminal Half-life (T1/2) of YKST02
Percentage of Participants with Anti-Drug Antibody (ADA) and Neutralizing Antibody (Nab) Against YKST02 | up to 42 weeks
  Assess the percentage of participants with ADA and Nab (only assessed when ADA positive) after treatment with YKST02.
ORR | From the date of dosing until the date of first documented progression
  Measured by IMWG criteria, only applicable in dose escalation phase
Progression-free Survival (PFS) | From the date of dosing until the date of first documented progression
  Evaluation of the efficacy of YKST02 in patients with MM on progression-free survival
Overall survival (OS) | From the date of first dose until loss of follow-up, death, withdrawal of informed consent, or the end of study, whichever occurs first
  Overall survival (OS) was defined as the time from the date of first dose until death due to any cause.
Minimal Residual Disease (MRD) Negativity Rate | From start of treatment to end of the study (approximately 42 weeks)
  MRD negativity rate was the percentage of participants with CR/sCR and negative MRD.

CONTACTS AND LOCATIONS:
Overall Officials: Wenming Chen, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (12):
- China (12):
  - Beijing Chao-yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Shunde Hospital of Southern Medical University, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanxi Cancer hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang